CLINICAL TRIAL: NCT06129682
Title: Self-rehabilitation At Home After LumbaR Arthrodesis
Brief Title: Self-rehabilitation At Home After LumbaR Arthrodesis (SAHARA)
Acronym: SAHARA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP230526; 2023-A00652-43 (Other: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Spondylolisthesis, Lumbar Region
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention)
- Self rehabilitation at home (Experimental)
  Interventions: Other: Self rehabilitation at home

INTERVENTIONS:
Other: Self rehabilitation at home — 6 week program of exercise at home of gradual intensity and duration
  Arms: Self rehabilitation at home

SUMMARY:
Lumbar arthrodesis is more and more common in general population. Patients need early reeducation after surgery but do not always have access to a physiotherapist.

The investigators aim to study the benefits of self-rehabilitation at home after lumbar arthrodesis, showing amelioration in lumbar pain and in quality of life for concerned patients. For this, the investigators designed a randomized-controlled study to test if self-rehabilitation at home right after surgery is superior than rehabilitation done by a physiotherapist 4 to 6 weeks after surgery (standard treatment for our patients).

DETAILED DESCRIPTION:
Due to population aging, lumbar arthrodesis is becoming more frequent in general population. At the same time, those patients need early rehabilitation, even if they do not experiment any motor disability after surgery : it has been showed that early rehabilitation improves lumbar pain thanks to muscle strengthening.

The design of the study is prospective,monocentric, controlled and randomized. This study compares progressive self-rehabilitation at home after lumbar arthrodesis, explained to the patient by a physiotherapist during his or her stay at the hospital and started right after surgery, versus rehabilitation done by a physiotherapist 4 to 6 weeks after surgery (standard treatment).

The primary outcome is decrease of lumbar pain at 6 weeks and 3 months after surgery. The secondary outcomes are improvement of functional abilities and improvement of pelvis and limbs ranges of motion.

Patients of both groups will be followed by surgeon and physiotherapist at 6 weeks and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar pain and/or nerve root pain and/or limp without any motor deficiency of the limbs, before and/or after surgery (if any motor deficiency occurs after surgery, it will be a secondary exclusion criteria)
* Surgery for posterolateral lumbar arthrodesis, from a degenerative etiology, from 1 to 3 lumbar levels (one level means one inter-somatic space)
* Surgery indication after optimal medical treatment, including appropriate pain medicine, and fail of medical treatment for reducing lumbar pain and/or nerve root pain and/or limp
* Return home possible after surgery
* After signing consent during pre-operative visit with the surgeon

Exclusion Criteria:

* People under 18 years-old
* Pregnant or breast-feeding women
* Psychiatric and/or neurodegenerative comorbidity
* Motor deficiency of the limbs before and/or after surgery
* Iliac extension of arthrodesis
* Any postoperative complication lengthening stay at hospital
* Medical contraindication for early rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change of lumbar pain | At 6 weeks and 3 months after surgery
  Improvement of Short Form 36 score (SF-36) Unit : number of points Each item is graded on a scale of 0 to 100, with 0 and 100 serving as the lowest and highest possible scores. A higher number indicates that the subject is in better overall health.

SECONDARY OUTCOMES:
Improvement of functional abilities | At 6 weeks and 3 months after surgery
  Improvement of Oswestry Disability Index (ODI) Unit : number of points The ODI consists of 10 patient-completed questions in which the response options are presented as 6-point Likert scales. Scores range from 0% (no disability) to 100% (most severe disability).
Improvement of ranges of motion - Ely test | At 6 weeks and 3 months after surgery
  Improvement of Ely test Angular unit : degree ( ° )
Improvement of ranges of motion - Straight Leg Test | At 6 weeks and 3 months after surgery
  Improvement of Straight Leg Test Angular unit : degree ( ° )
Improvement of ranges of motion - Schober test | At 6 weeks and 3 months after surgery
  Improvement of Schober test angular unit : degree ( ° )

CONTACTS AND LOCATIONS:
Overall Officials: Marc Khalifé, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP - Hôpital Européen Georges-Pompidou Paris, France, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).